CLINICAL TRIAL: NCT06128915
Title: The Role of Neutrophils in the Age-driven Decline in Anti-pneumococcal Vaccine Responses
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Elsa Bou Ghanem, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00007111; R01AG068568 (NIH)
Record Dates: First submitted 2023-10-30; First posted 2023-11-13 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Aging
Keywords: Aging; Neutrophils; Streptococcus pneumoniae; Pneumococcal conjugate vaccine
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: Vaccination with Prevnar.
Masking Description: Enrolled participants will be assigned a unique study identification number followed by a visit number (example 1.1 for donor #1-first visit). The code list, linking patient identities (such as names/phone numbers) and samples, will be kept in a separate file locked in a drawer the PI's office. The code list and code-identified data will be stored in separate locations and only authorized individuals will have access to the list. Experiments and data analysis will be performed only on coded samples and researchers will only have access to the visit number as the experiments to be performed on the collected samples pre and post vaccination differ.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vaccination with Prevnar. (Experimental): Intramuscular vaccination with Prevnar 20
  Interventions: Other: vaccine

INTERVENTIONS:
Other: vaccine — Vaccination against 20 serotypes of S. pneumoniae

SUMMARY:
This study focuses on the role of neutrophils in shaping the adaptive immune response to the anti-pneumococcal vaccine Prevnar-13 in young and elderly adults.

DETAILED DESCRIPTION:
This study focuses on the role of neutrophils in shaping the adaptive immune response to the anti-pneumococcal vaccine Prevnar in young and elderly adults. This study involves direct vaccination of human volunteers. The endpoints will be determining how vaccination affects neutrophil responses and linking those neutrophil responses to antibody responses following vaccination. The main results will be:

1. Elucidating how neutrophils kill bacteria before and after vaccination
2. Elucidate the phenotype of neutrophils before and after vaccination
3. Elucidate how neutrophils interact with B and T cell in vitro before and after vaccination
4. Measure antibody levels and function before and after vaccination
5. Correlate neutrophil responses to antibody levels and function

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Have not been vaccinated with any licensed or experimental pneumococcal vaccine
* Ages 21-40; and ≥65. Individuals >60 years old will also be recruited in case we find no unvaccinated people ≥65 years old
* Free of acute infections within the last 2 weeks
* Did not take any anti-inflammatory medicine in the last week
* Did not ingest alcohol in the last 24 hours
* Ability and willingness to provide consent

Exclusion Criteria:

* Previous vaccination with any licensed or experimental pneumococcal vaccine
* Known hypersensitivity to vaccination and vaccine components
* Immune deficiency
* Use of immune-modulating or suppressive drugs
* Malignancies within the last 2 years
* Known hematological, rheumatic and inflammatory diseases
* Known chronic infections
* Poorly controlled chronic cardiovascular and metabolic conditions
* Pregnancy
* Dementia

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Pneumococcal Opsonophagocytic Killing Activity (OPH) by neutrophils from young versus old donors at 1 week and 1 month after vaccination | 1 month
  OPH will be determined by measuring the percentage of S. pneumoniae bacteria killed in vitro by neutrophils from donors

SECONDARY OUTCOMES:
Surface phenotype of neutrophils from young versus old donors at 1 week and 1 month after vaccination | 1 month
  Phenotype will be determined by measuring the expression of surface receptors on neutrophils ex vivo by flowcytometry from donors

CONTACTS AND LOCATIONS:
Overall Officials: Elsa N Bou Ghanem, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No